CLINICAL TRIAL: NCT01570322
Title: Determinants of Quality of Life Related to Health in Alzheimer Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PN09004
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Alzheimer Disease
Keywords: Dementia - Alzheimer - Quality of life
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study the factors that explain Health-Related Quality of Life (HRQL) in patients with Alzheimer disease including:

* The influence of the environment (physical and human) on Health-Related Quality of Life (HRQL),
* The influence of non-drug and drug treatments on Health-Related Quality of Life (HRQL),
* The influence of formal and informal help mobilized,
* The influence of interactions "patient - caregiver" on Health-Related Quality of Life (HRQL),
* The influence of the ratio necessary cost on available resources on Health-Related Quality of Life (HRQL)

ELIGIBILITY:
Inclusion Criteria:

* Patients with Alzheimer disease (DSM IV and NINCDS-ADRDA)
* Patients with MMSE (Mini Mental State Examination) > or = 10
* Out patients

Exclusion Criteria:

* Severe sensory disturbances,
* Non French speaking

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: * Patients with Alzheimer disease (DSM IV - Diagnostic and Statistical Manual of Mental Disorders - and NINCDS/ADRDA - National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association)
  * Patients with MMSE (Mini Mental State Examination) > or = 10
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQOL) Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de REIMS, Reims, France, France